CLINICAL TRIAL: NCT03143673
Title: ACURATE™ Transapical Aortic Bioprosthesis for Implantation in Patients With Severe Aortic Stenosis
Brief Title: ACURATE™ Transapical Aortic Bioprosthesis for Implantation in Patients With Severe Aortic Stenosis (2010-01)
Acronym: TA-PILOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-01; 95.02-5660-6278 (Other: Bundesinstitut für Arzneimittel und Medizinprodukte (BfArM))
Record Dates: First submitted 2014-12-08; First posted 2017-05-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Aortic Symptomatic Stenosis
Keywords: Severe Symptomatic Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACURATE TA™ (Experimental): Patient implanted with ACURATE TA™ Bioprosthesis
  Interventions: Device: ACURATE TA™

INTERVENTIONS:
Device: ACURATE TA™ — ACURATE TA™ Transapical Aortic Bioprosthesis is intended for subjects with severe symptomatic Aortic Stenosis and are considered high risk for surgical conventional Aortic Valve Replacement Surgery.
  Other Names: ACURATE TA™ Transapical Aortic Bioprosthesis and Delivery System

SUMMARY:
The purpose of this study is to evaluate safety of the study device and study device performance in patients presenting with severe aortic stenosis who are considered to be high risk for open surgical repair.

DETAILED DESCRIPTION:
A single arm, prospective, multicenter, non-randomized, and open trial, up to 5 years follow-up with the Symetis ACURATE TA™ which is an aortic bioprosthesis for minimal invasive implantation vie transapical access to treat patients with severe symptomatic aortic stenosis where conventional aortic valve replacement (AVR) via open heart surgery is considered to be associated with high surgical risk for evaluating safety and performance of the implantation and safety at 30-D follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 75 years of age
2. Additive EuroSCORE > 9
3. Severe AS assessed by echocardiography and documented by a mean gradient > 40mmHg and a native Aortic Valve Area (AVA) < 0.8 cm² or Aortic Valve Area Index (AVAI) < 0.6 cm²/m²
4. NYHA Functional Class > II
5. Aortic annulus (AAn) diameters between and including 21 mm up to 27 mm (21mm ≤ AAn ≤27mm) by transoesophageal echocardiography (TEE)
6. Patient understands the implications of participating in the study and provides signed informed consent

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve
2. Severe eccentricity of calcification
3. Severe mitral regurgitation (> 2°)
4. Pre-existing prosthetic heart valve in any position and / or prosthetic ring
5. Severe transapical access problem, non-reachable LV apex
6. Previous surgery of the LV using a patch, such as the Dor procedure
7. Presence of apical LV thrombus
8. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
9. Acute myocardial infarction (AMI) within 1 month prior to the procedure
10. PCI within 1 month prior to the procedure
11. Previous transient ischemic attack (TIA) or stroke in the last 3 months
12. Untreated clinically significant coronary artery disease (CAD) requiring revascularization
13. Hemodynamic instability: systolic pressure <90mmHg without afterload reduction, shock, need for inotropic support or intra-aortic balloon pump
14. Severe left ventricular dysfunction (LVEF) < 30% by echocardiography
15. Calcified pericardium
16. Septal hypertrophy unacceptable for transapical procedure
17. Primary hypertrophic obstructive cardiomyopathy (HOCM)
18. Active infection, endocarditis or pyrexia
19. Active peptic ulcer or gastrointestinal (GI) bleeding within the past 3 months
20. Significant hepatic involvement (Child > B)
21. Severe COPD requiring home oxygen
22. History of bleeding diathesis or coagulopathy
23. Hematologic disorder (WBC < 3000mm3, Hb < 9g/dL, platelet count < 50000 cells/ mm3)
24. Chronic renal dysfunction with a serum creatinine level > 2.5 mg/dL or renal failure requiring dialysis
25. Neurological disease severely affecting ambulation or daily functioning, including dementia
26. Another surgical or percutaneous procedure scheduled at the same time
27. Emergency procedure
28. Life expectancy < 12 months due to non-cardiac co-morbid conditions
29. Known hypersensitivity/contraindication to any study medication, contrast media, or nitinol
30. Currently participating in an investigational drug or another device study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Freedom from all-cause mortality at 30 day Follow Up | 30-Day Follow-up
  The primary study objective is to evaluate the safety of the ACURATE™ Transapical Aortic Bioprosthesis at 30 days post-procedure in patients presenting with severe aortic valve stenosis at high risk for conventional AVR surgery.
Freedom from all-cause mortality at 12 months Follow Up | 12 months Follow-Up
  The primary study objective is to evaluate the safety of the ACURATE™ Transapical Aortic Bioprosthesis at 12 months post-procedure in patients presenting with severe aortic valve stenosis at high risk for conventional AVR surgery.

SECONDARY OUTCOMES:
Rate of Major Adverse Valve-Related Events (MAVRE) at 30 days and at 12 month follow up related to the study device as defined as; | 30-Days and at 12 Months Follow-up
  2.1 Structural valve deterioration
  2.2 Non-structural dysfunction of the implanted study device
  2.3 Valve thrombosis, embolism, bleeding event
  2.4 Operated valve endocarditis
  2.5 Re-intervention on the implanted device
  2.6 Valve-related mortality
  2.7 Need for new permanent pacemaker or defibrillator within 14 days
Rate of Major Adverse Cardiac and Cerebrovascular-Related Events (MACCE) at 30 days and at 12 Month and defined as cardiovascular death, myocardial infarction and stroke. | 30-Day and 12-Month
  Defined as cardiovascular death, myocardial infarction and stroke
Functional Improvement from baseline | 30-Days and 12-Month Follow-up
  per NYHA functional classification
Procedural success | 24 hours Post-Procedure
  defined as stable study device placement at intended site and adequate device functioning immediately post-implantation, confirmed by angiography and echocardiography as assessed at a Core Lab and without intraprocedural mortality.
Device success at 30 Days and 12 Month follow-up as defined as adequate functioning of the study device as confirmed by angiography and/or echocardiography as assessed at a CoreLab. | 30-Day and 12-Month Follow-up
  Device success at 30 Days and 12 Month follow-up as defined as adequate functioning of the study device as confirmed by angiography and/or echocardiography as assessed at a CoreLab. The following datapoints will be analyzed:
  6.1 Effective orifice area and index (EOA/EOAI)
  6.2 Transvalvular Gradients (Peak and mean)
  6.3 Paravalvular and intravalvular (Central) leaks
  6.4 Aortic Insufficiency
  6.5 LV function and hemodynamics
  6.6 Valve function and morphology

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walther, Professor, Principal Investigator — Kerckhoff Klinik
Locations (5):
- Germany (5):
  - Kerckhoff Klinik GmbH, Bad Nauheim
  - Universitätsklinikum Hamburg-Eppendorf Klinik für Herz-und Gefässchirurgie, Essen
  - Universitätsklinikum Essen Westdeutsches Herzzentrum Essen, Essen
  - Klinik für Herzchirurgie GmbH, Karlsruhe
  - Herzzentrum Leipzig GmbH, Leipzig